CLINICAL TRIAL: NCT05278117
Title: A Prospective Multicentre Study Evaluating the Outcomes of the Abdominal Wall Dehiscence Repair Using Posterior Component Separation With Transversus Abdominis Muscle Release Reinforced by a Retro-muscular Mesh - Filling a Step
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, assistant professour of general and laparoscopic surgery, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: burst abdomen
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Abdominal Wall Defect
Keywords: Abdomen burst, Incisional hernia, mesh
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- complete burst abdomen repair (Experimental): complete burst abdomen repair
  Interventions: Procedure: outcomes of complete burst abdomen repair using posterior component separation technique with transversus abdominis muscle release reinforced by sublay mesh

INTERVENTIONS:
Procedure: outcomes of complete burst abdomen repair using posterior component separation technique with transversus abdominis muscle release reinforced by sublay mesh — outcomes of complete burst abdomen repair using posterior component separation technique with transversus abdominis muscle release reinforced by sublay mesh

SUMMARY:
Purpose: This study determined the incidence of burst abdomen recurrent (BAR), incisional hernia(IH), and surgical site occurrence (SSO) following burst abdomen surgical treatment after abdominal midline incisions using a posterior component separation(CS) technique with transversus abdominis muscle release (TAR) reinforced by retro-muscular mesh technique.

Methods: Between June 2014 and April 2018, 202 patients with grade IA BA (Björck's first classification) were treated in a prospective multiple-center cohort study.

DETAILED DESCRIPTION:
This study determined the incidence of burst abdomen recurrent (BAR), incisional hernia(IH), and surgical site occurrence (SSO) following burst abdomen surgical treatment after abdominal midline incisions using a posterior component separation(CS) technique with transversus abdominis muscle release (TAR) reinforced by retro-muscular mesh technique.

Methods: Between June 2014 and April 2018, 202 patients with grade IA BA (Björck's first classification) were treated in a prospective multiple-center cohort study.

ELIGIBILITY:
Inclusion Criteria:

* BA Grade IA according to Björck's initial classification following midline laparotomy from various departments,
* ≥ 18 years
* both sex
* emergency or elective surgery

Exclusion Criteria:

* BA grade 1B,2,3, and 4 according to Björck's initial classification,
* < 18 years,
* primary laparotomy performed through a non-midline incision, open abdomen,
* if another laparotomy had been performed between the surgery for BA and the end of the follow-up period,
* concomitant intra-abdominal surgery, abdominal complications during BA surgery,
* adherent bowel to the defect edge that cannot be separated,
* patients lost during follow up,
* presence of intra-abdominal contamination that cannot be controlled radiologically,
* history of previous BA repair,
* stoma exteriorized from the midline primary wound,
* temporarily wound closure techniques,
* prior abdominal surgeries other than operation resulted in BA,
* prior abdominal wall hernia repair with or without mesh,
* history of collagen diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
recurrent burst abdomen | 3.5 years
  incidence of recurrent burst abdomen by %
incisional hernia | 3.5 years
  incidence of incisional hernia measured by clinical examination and computerized tomography by %

SECONDARY OUTCOMES:
incidence of surgical site infection | 30 days
  by %

CONTACTS AND LOCATIONS:
Overall Officials: Alnaimy alnaimy, Phd, Principal Investigator — Zagazig University
Locations (1):
- Tamer Alsaied Alnaimy, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Habeeb TAAM, Hussain A, Shelat V, Chiaretti M, Bueno-Lledo J, Garcia Fadrique A, Kalmoush AE, Elnemr M, Safwat K, Raafat A, Wasefy T, Heggy IA, Osman G, Abdelhady WA, Mawla WA, Fiad AA, Elaidy MM, Amr W, Abdelhamid MI, Abdou AM, Ibrahim AIA, Baghdadi MA. A prospective multicentre study evaluating the outcomes of the abdominal wall dehiscence repair using posterior component separation with transversus abdominis muscle release reinforced by a retro-muscular mesh: filling a step. World J Emerg Surg. 2023 Mar 3;18(1):15. doi: 10.1186/s13017-023-00485-9. PMID 36869364